CLINICAL TRIAL: NCT02004899
Title: Onset of Labor Epidural Analgesia With Low Dose Bupivacaine and Different Doses of Fentanyl: a Randomized Double Blinded Clinical Trial.
Brief Title: Trial of Onset of Epidural Pain Relief With Low Dose Bupivacaine and Different Doses of Fentanyl in Laboring Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Indu Singh, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 104456
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Anesthetic, Sedative or Analgesic Complications in Labor or Delivery
Keywords: Labor epidural analgesia; Fentanyl; Bupivacaine; Onset
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- F20 (Active Comparator): Patients randomized to this arm of the study receive 20 mcg fentanyl and 8 mg bupivacaine as their epidural loading dose
  Interventions: Drug: Fentanyl
- F50 (Experimental): Patients randomized to this arm of the study receive 50 mcg fentanyl with 8 mg bupivacaine as their epidural loading dose
  Interventions: Drug: Fentanyl
- F100 (Experimental): Patients randomized to this arm of the study receive 100 mcg fentanyl and 8 mg bupivacaine as their epidural loading dose
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — After obtaining informed consent, patients are randomized into one of two treatment groups or a control group by a computer generated random number table. After confirmation of epidural placement following test dose administration, a loading dose of 10 ml 0.08% Bupivacaine containing 20 mcg Fentanyl is administered after adding 1.6 ml 0.9% NaCl (Sodium Chloride) in the control group (F20).
  Other Names: Duragesic, Actiq

SUMMARY:
Epidural analgesia is the most effective form of labor pain relief. Low doses of local anesthetic (freezing solutions) in combination with opioids (narcotics) are commonly used as epidural solutions to provide pain relief. Low dose local anesthetic solutions with opioids for labor have been shown to decrease motor block (leg weakness or temporary paralysis), without affecting labor pain relief. However, onset of pain relief can be delayed with these low dose solutions. The standard epidural solution used at Victoria Hospital is a low dose of local anesthetic called bupivacaine mixed with fentanyl, an opioid, for labor epidural pain relief.

There is some evidence that the addition of more fentanyl to the epidural bolus dose of bupivacaine at the start of labor epidural analgesia can speed onset of pain relief. Both medications are safe for you and your baby.

This study will investigate whether the addition of different doses of fentanyl (20 mcg, 50 mcg and 100 mcg) to the epidural bolus dose speeds onset of pain relief.

The study hypothesis is that the onset of epidural labor analgesia will be shortest with the larger fentanyl epidural bolus.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 or 2
* Pregnant women in early labor (cervical dilation <5cm)
* Singleton fetuses
* Gestational age more than 36 weeks
* Normal fetal heart rate tracing

Exclusion Criteria:

* Severe pre-ecclampsia
* Antepartum hemorrhage
* ASA >3
* Chronic pain
* Substance abuse
* Language barrier between patient and investigator
* Contraindications to epidural analgesia
* Allergies to local anesthetics or fentanyl
* Morbid obesity
* Previous administration of opioid analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The time, in minutes, since completion of epidural bolus to the first painless contraction | Time since epidural bolus dose administration (At 1 and 5 minutes )
  A painless contraction = verbal Numeric Pain Rating Scale less than or equal to 3/10

SECONDARY OUTCOMES:
Sensory block height to ice | 30 minutes after epidural bolus dose
Pruritis | 30 minutes after epidural bolus dose
  Pruritus will be measured using a 4-point scale, where 0 is none, 1 is mild, 2 is moderate, and 3 is severe.
Nausea | 30 minutes after epidural bolus dose
  Nausea will be measured using a 4-point scale, where 0 is none, 1 is mild, 2 is moderate, and 3 is severe.
Maternal sedation | 30 minutes after epidural bolus dose
  Maternal sedation will be measured using a 5-point scale where 0 is wide awake, 1 is mildly drowsy, 2 is very drowsy, 3 is asleep but rousable, and 4 is somnolent.
Hypotension | 30 minutes after epidural bolus dose
  Hypotension is defined as a decrease in systolic blood pressure by 30% or more, or less than 90 mmHg. It is treated with intravenous ephedrine.
Motor block | 30 minutes after epidural bolus dose
  Motor block will be assessed using a modified Bromage score (0 = ability to move hips, ankles, and knees, 1 = inability to raise extended leg, 2 = inability to flex knee, and 3 = inability to flex ankle, foot or knee).
Time, in minutes, from epidural bolus dose to use of patient controlled epidural demand dose | Estimated time frame 1 hour
  time after epidural loading dose at which patient uses Patient Controlled Epidural Analgesia administered bolus
Patient satisfaction of analgesia | 30 minutes from epidural bolus dose
  Patient satisfaction of analgesia will be measured using a 5-point scale where 0 is completely dissatisfied, 1 is somewhat dissatisfied, 2 is neutral, 3 is somewhat satisfied, and 4 is completely satisfied.
Incidence of failed analgesia | 30 minutes after epidural bolus dose
  Patients who have a verbal Numeric Rating Scale score greater than 3/10 after 30 minutes of epidural bolus dose will be deemed a failure.
Incidence of fetal bradycardia | Estimated time frame 24 hours
Time, in minutes, from completion of epidural test dose to delivery | Estimated time frame 24 hours
Type of delivery | Estimated time frame 24 hours
Fetal birth weight | Estimated time frame 24 hours
Neonatal Apgar scores | At 1 and 5 minutes post-delivery
Breastfeeding | 24 hours after delivery
  Has breastfeeding been established at 24 hours post-delivery?

CONTACTS AND LOCATIONS:
Overall Officials: Indu Singh, Principal Investigator — Schulich School of Medicine and Dentistry/Anaesthesia
Locations (1):
- Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available